CLINICAL TRIAL: NCT02353065
Title: Sonographic Assessment of Reduction in Colles' Fracture
Acronym: SONAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simon Richards (Other)
Collaborators: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Simon Richards, Senior Lecturer Medical Imaging (Ultrasound), Teesside University
Organization: Teesside University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 141/13
Record Dates: First submitted 2015-01-25; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Colles' Fracture
Keywords: Colles' Fracture; ultrasonography
MeSH Terms: conditions — Colles' Fracture | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Assessment of adequacy of reduction by bedside x-ray during period of intravenous regional anaesthesia (Biers block)
  Interventions: Radiation: Bedside x-ray
- Ultrasound (Experimental): Assessment of adequacy of reduction by bedside ultrasound performed by the treating clinician during period of intravenous regional anaesthesia (Biers block)
  Interventions: Procedure: Ultrasound imaging

INTERVENTIONS:
Procedure: Ultrasound imaging — Point of care ultrasound of fracture site during and post-reduction
  Arms: Ultrasound
Radiation: Bedside x-ray — Portable x-ray of fracture post-reduction
  Arms: Control

SUMMARY:
Colles fractures are a common type of wrist fracture that often requires manipulation in the Emergency Department. Currently xrays are used to assess whether this has been successful, which are done once the plaster cast has been applied. This study will assess whether ultrasound can be used immediately after the manipulation to check the position, before the plaster cast is applied. This would then be followed by an xray as normal.

The aim is to assess the feasibility of a full study to determine which method is faster, causes less pain, and also to assess if either approach reduces the need for repeat attempts at manipulation and surgical repair.

DETAILED DESCRIPTION:
Fractures of the distal radius are a frequent cause for presentation to United Kingdom (UK) Emergency Departments, and the Colles' fracture is the most commonly encountered type. These injuries frequently occur in isolation, or associated with only minor injuries, and reduction of displaced fractures is typically performed by Emergency Physicians at the time of first attendance to the hospital.

The usually sequence of events is clinical examination, x-ray imaging to confirm the fracture, then the reduction is performed with appropriate analgesia or anaesthesia, the arm placed in a plaster backslab, and repeat imaging is taken to confirm adequacy of reduction. If the reduction is not satisfactory, repeat manipulation is required.

Haematoma block and Biers block permit x-ray imaging of the manipulated wrist while the anaesthetic action is still effective, permitting re-manipulation without further administration of local anaesthetic. Sedation is usually kept to as short a time as possible, and is not usually maintained while imaging is performed. There is usually some degree of delay while x-rays are taken and made available for viewing, and this wait prolongs the procedure for the patient and the treating clinician. In addition, Biers block cannot be tolerated for long by most patients, so any delay makes it less likely that a re-manipulation can be achieved within the time the patient can tolerate. If a patient has been sedated, a re-manipulation will require a further sedative (or alternative) procedure with the concomitant risks that entails.

Ideally, imaging would be performed rapidly, immediately at the end of the manipulation, prior to application of plaster, allowing confirmation of the reduction or immediate re-manipulation if necessary. This description of imaging provided at the point of care by the treating clinician, aimed at answering a clearly defined question ('is this an adequate reduction?') matches the description of focussed emergency ultrasound in other applications. If ultrasound could be used to assess fracture reduction, it would have potential to save clinician time, patient time and discomfort, and reduced the need for repeated manipulations and surgical repair.

This study intends to assess the feasibility of a full trial of efficacy comparing ultrasound with x-ray to guide the reduction of these fractures.

ELIGIBILITY:
Inclusion Criteria:

* Adults with isolated fractures of the distal radius undergoing manipulation in the Emergency Department with Intravenous Regional Anaesthesia (Biers Block)

Exclusion Criteria:

* Age under 16
* Contraindication to Biers block
* Unable to give informed consent
* Multiple injuries
* Open fracture
* Prisoners

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The total inflation time of the tourniquet used during the Biers Block | The duration the tourniquet is inflated; complete within 30 minutes of the procedure commencing
  The total inflation time of tourniquet used for Biers block

SECONDARY OUTCOMES:
The total number of manipulations required per patient within the Emergency Department | The duration of the manipulation procedure; complete within 30 minutes of procedure commencing
  Number of attempts at manipulation within Emergency Department
Does the use of ultrasound reduce the need for surgical reduction? | Four weeks from visit
  Need for surgical reduction/fixation
Does the use of ultrasound reduce the time spent within the Emergency Department? | End of initial ED visit, within twelve hours of initial arrival to the hospital
  Total time spent within Emergency Department
Does the use of ultrasound reduce the pain score during the reduction? | End of procedure - within 30 minutes of the procedure commencing
  Patient reported pain score at the end of the fracture reduction
Does the use of ultrasound increase the patient satisfaction? | Four weeks after visit
  Patient reported satisfaction with reduction of fracture

CONTACTS AND LOCATIONS:
Overall Officials: Simon Richards, Principal Investigator — Teesside University
Locations (1):
- Royal Preston Hospital, Preston, Lancashire, United Kingdom